CLINICAL TRIAL: NCT04592250
Title: Financial Toxicity in Diverse Cancer Populations and Care Settings
Brief Title: Financial Toxicity in Cancer Patients
Status: Active, not recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2020-0356; NCI-2020-07501 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0356 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-10-12; First posted 2020-10-19 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational (survey): Participants will complete a survey packet that is estimated to take about 30 minutes. The survey packet will be collected at baseline and at 6 months.
  Interventions: Other: Survey Administration

INTERVENTIONS:
Other: Survey Administration — Complete survey

SUMMARY:
This study will seek to generate the early data needed to understand the relationship between constructs and measures of patients' coping resources and psychological response and measures of patients' financial toxicity. To collect this early descriptive data, the overall goal of this study is to identify social, behavioral, and knowledge factors associated with financial toxicity outcomes. Identifying these factors will ultimately help elucidate targets for behavioral, psychosocial, and/or educational and coaching interventions.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

1. Examine the associations between measures of self-efficacy, quality of social support, and financial literacy with the outcome measure of financial toxicity.
2. Identify the feasibility of collecting these measures in a Spanish-speaking cancer patient population.
3. Describe the relationship between financial toxicity and clinical outcomes (survival and disease status). This is an exploratory aim.
4. a) Describe the correlation between measures of self-efficacy, quality of social support, financial literacy and clinical and demographic patient characteristics with outcome measure of financial toxicity, by tumor type and age subgroups. b) Describe response rate to the financial toxicity measure (>50% completed items on the survey instrument), by tumor type and age subgroups. This is an exploratory aim.

OUTLINE:

Participants will complete a survey packet that is estimated to take about 30 minutes. The survey packet will be collected at baseline and at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be able to read and speak English or Spanish
* Participant must have diagnosis of cancer within the past 365 days; all disease sites and all stages are eligible for enrollment

Exclusion Criteria:

* Unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who have a diagnosis of cancer within the past 365 days
Sampling Method: Non-Probability Sample
Enrollment: 625 (Estimated)
Dates: Start 2020-09-12 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Financial toxicity score | At 6 months
  Will be measured using the ENRICh instrument. Will conduct descriptive and univariate/multivariate analyses on this association of primary interest, including Chi-square test, t-test (or non-parametric test as appropriate). Other univariate associations between financial toxicity and other covariates obtained from survey measures, considered descriptive, will be performed. will test the primary association between the Hope State measure and financial toxicity using multivariate generalized linear mixed models, accounting for longitudinal changes in outcome scores over time, as well as adjusting for covariates and potential time interactions. The mixed effects structure will also be used, via a random intercept term, to account for site-to-site differences (e.g. clustering). Standard model selection procedures (forward, backward, or stepwise selection or shrinkage penalty) will be applied to determine the final multivariate model.

CONTACTS AND LOCATIONS:
Overall Officials: Grace Smith, Principal Investigator — M.D. Anderson Cancer Center
Locations (6):
- United States (6):
  - DCH Regional Medical Center, Tuscaloosa, Alabama
  - Scripps - MD Anderson Cancer Center, La Jolla, California
  - Baptist- MD Anderson Cancer Center, Jacksonville, Florida
  - The Queen's Medical Center, Honolulu, Hawaii
  - Lyndon Baines Johnson General Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center — http://www.mdanderson.org